CLINICAL TRIAL: NCT06634212
Title: Validity and Reliability of Dubousset Functional Test in Total Knee Arthloplasty
Brief Title: The Dubousset Functional Test in Total Knee Arthloplasty
Acronym: DFT-TKA
Status: Not yet recruiting | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Asistant Professor, Physiotherapist, Alanya Alaaddin Keykubat University
Other Study IDs: 2024/DFT-TKA
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and reliability of Dubousset Functional Test in the patients with Total Knee Prothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had Total Knee Arthroplasty
* Patients aged 50-70 years.

Exclusion Criteria:

* Patients who didn't have any Total Kne arthroplasty
* hose with fractures, pregnancy, a disease that would prevent physical exertion, those with a body mass index (BMI) of 40 kg/m2 and above, and those with major musculoskeletal or neurological disorders that cause gait disturbance will be excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-70 years who had Total Knee Arthroplasty
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Dubousset Functional Test | 10 minutes
  The four test components included the Up and Walking Test (unassisted sit-to-stand from a chair, walk forward/backward 5 meters [no turn], then unassisted stand-to-sit), Steps Test (ascend three steps, turn, descend three steps), Down and Sitting Test (stand-to-ground, followed by ground-to-stand, with assistance as needed), and Dual-Tasking Test (walk 5 meters forwards and back while counting down from 50 by 2).

IPD SHARING:
Plan to Share IPD: No